CLINICAL TRIAL: NCT07168109
Title: Visual Outcomes of an Enhanced Monofocal Intraocular Lens Targeted for Monovision in Highly Myopic Eyes: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Shenzhen Eye Hospital (Other)
Responsible Party: Principal Investigator, Lixia Luo, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KYPJ072
Record Dates: First submitted 2025-09-02; First posted 2025-09-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Cataract; High Myopia
Keywords: high myopia; cataract; impaired visual acuity
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monovision group (Experimental): Both eyes will be implanted with enhanced monofocal intraocular lenses, with the dominant eye targeted for -0.5 diopters (D) and the nondominant eye for -2.0 D.
  Interventions: Procedure: Enhanced monofocal intraocular lens implantation (monovision strategy)
- Bilateral myopia group (Active Comparator): Both eyes will be implanted with enhanced monofocal intraocular lenses, with each eye targeted for -2.0 D.
  Interventions: Procedure: Enhanced monofocal intraocular lens implantation (bilateral myopia strategy)

INTERVENTIONS:
Procedure: Enhanced monofocal intraocular lens implantation (monovision strategy) — Participants will undergo phacoemulsification with the implantation of an enhanced monofocal intraocular lens, targeting -0.5 D in the dominant eye and -2.0 D in the non-dominant eye. The first operated eye will be selected based on the worse corrected distance visual acuity; if both eyes are similar, the eye subjectively perceived by the patient as having worse vision will be chosen. The second eye surgery will be performed within 2 weeks after the first eye surgery. Ocular dominance will be determined preoperatively using the "finger method" . Intraocular lens power will be calculated using multiple formulas [Emmetropia Verifying Optical (EVO) version 2.0, Kane, LISA].
  Arms: Monovision group
Procedure: Enhanced monofocal intraocular lens implantation (bilateral myopia strategy) — Participants will undergo phacoemulsification with the implantation of an enhanced monofocal intraocular lens, targeting -2.0 D in both eyes. The first operated eye will be selected based on the worse corrected distance visual acuity; if both eyes are similar, the eye subjectively perceived by the patient as having worse vision will be chosen. The second eye surgery will be performed within 2 weeks after the first eye surgery. Ocular dominance will be determined preoperatively using the "finger method". Intraocular lens power will be calculated using multiple formulas [Emmetropia Verifying Optical (EVO) version 2.0, Kane, LISA].
  Arms: Bilateral myopia group

SUMMARY:
The goal of this clinical trial is to evaluate whether an enhanced monofocal intraocular lens targeted for monovision can improve visual outcomes in patients with cataract and high myopia (axial length ≥ 26 mm).

The main questions it aims to answer are:

For people with cataract and high myopia, does an enhanced monofocal intraocular lens targeted for monovision provide greater binocular uncorrected distance visual acuity compared with targeting myopia in both eyes? Does an enhanced monofocal intraocular lens targeted for monovision provide comparable binocular uncorrected intermediate and near visual acuity, contrast sensitivity, reading ability, spectacle independence, stereopsis, and photic phenomena compared with targeting myopia in both eyes?

Researchers will compare an enhanced monofocal intraocular lens targeted for monovision with one targeted for myopia in both eyes to determine whether the monovision strategy is more effective.

Participants will:

Undergo phacoemulsification with enhanced monofocal intraocular lens implantation. Attend follow-up visits at 1, 3, 6, and 12 months after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years (inclusive), no gender restrictions;
2. Scheduled to undergo bilateral phacoemulsification with intraocular lens implantation;
3. Axial length ≥ 26.0 mm in both eyes;
4. Desire for postoperative spectacle independence;
5. Able to understand and cooperate with the trial procedures, voluntarily participate in this clinical trial, and sign an informed consent form.

Exclusion Criteria:

1. Poor-quality preoperative ocular biometry (Axial length, keratometry, anterior chamber depth);
2. Preoperative corneal astigmatism ≥ 1.5 diopters (D);
3. Patients with intraoperative or postoperative complications (ie, intraoperative posterior capsular rupture, zonular dehiscence, secondary glaucoma, etc.);
4. The presence of other ocular diseases (ie, strabismus, severe retinal pathology, uveitis, other relevant ophthalmic diseases that might affect outcomes or trauma, etc.);
5. A history of intraocular surgery;
6. Severe chronic systemic diseases, psychiatric disorders, dementia, hearing impairments, or mobility limitations that would interfere with understanding of the monovision design, attendance at follow-up visits, or completion of questionnaires.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Binocular uncorrected distance visual acuity at 4 m | 3 months (±2 weeks) following the second eye surgery
  measured by the ETDRS chart

SECONDARY OUTCOMES:
Monocular and binocular uncorrected distance visual acuity at 4 m | 1, 6, 12 months following the second eye surgery
  measured by the ETDRS chart
Monocular and binocular uncorrected intermediate visual acuity at 80cm and 60cm | 1, 3, 6, 12 months following the second eye surgery
  measured by the EDTRS chart
Monocular and binocular uncorrected near visual acuity at 40cm | 1, 3, 6, 12 months following the second eye surgery
  measured by the EDTRS chart
Monocular and binocular defocus curves | 3, 6, 12 months following the second eye surgery
  measured by the binoptometer 4P
Stereoscopic vision | 3, 6, 12 months following the second eye surgery
Patient-reported outcome measures (PROMs): Vision-specific quality of life | 3, 6, 12 months following the second eye surgery
  Vision-specific quality of life is measured by the Chinese version of the 9-item short-form of the Catquest questionnaire (Catquest-9SF). There are five text response options for the answers, scaled from "Yes, very great difficulties" to "No, no difficulties", including the answer "Cannot decide". The minimum score is 9, and the maximum score is 36.
Patient-reported outcome measures (PROMs): Photic phenomena | 3, 6, 12 months following the second eye surgery
  Pictures from the Quality of Vision (QoV) questionnaire were shown to patients, who were then asked to rate the frequency (never, occasionally, quite often, very often), severity (none, mild, moderate, severe) of photic phenomena and the extent to which these phenomena interfered with daily life (not at all, a little, quite, very).
Patient-reported outcome measures (PROMs): Spectacle independence | 3, 6, 12 months following the second eye surgery
  Spectacle independence is measured by a self-made spectacle independence questionnaire. Patients will be asked about the frequency of spectacle independence at the distance, intermediate, and near distances. There are three text response options for the answers, including "Always", "Seldom", and "Never".

OTHER OUTCOMES:
Binocular contrast sensitivity | 3, 6, 12 months following the second eye surgery
Reading ability | 3, 6, 12 months following the second eye surgery
  measured by the International Reading Speed Texts (IResT)
Intraoperative or postoperative complications | 1, 3, 6, 12 months following the second eye surgery
  Clinical manifestations are assessed and recorded by the ophthalmologist.
Self-reported incidence and severity of ocular discomfort | 1, 3, 6, 12 months following the second eye surgery
  collected by self-reported outcomes and past medical records (if any) of participants